CLINICAL TRIAL: NCT06717360
Title: A Multicenter, Randomized, Double-blinded, Active-controlled, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of AG2304T and AG2304R in Patients with Primary Hypercholesterolemia
Brief Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of AG2304T and AG2304R
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG2304 P3
Record Dates: First submitted 2024-11-28; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AG2304T (Experimental)
  Interventions: Drug: AG2304T
- AG2304R (Active Comparator)
  Interventions: Drug: AG2304R

INTERVENTIONS:
Drug: AG2304T — AG2304T, QD, PO
  Arms: AG2304T
Drug: AG2304R — AG2304R, QD, PO
  Arms: AG2304R

SUMMARY:
A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of AG2304T and AG2304R in Patients with Primary Hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19-80
* Patients with primary hypercholesterolemia
* Those who voluntarily written consent to participate in this clinical trial

Exclusion Criteria:

* The subject not meet the specified LDL-C level
* Other exclusions applied

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
LDL-C level | 8 weeks

IPD SHARING:
Plan to Share IPD: No